CLINICAL TRIAL: NCT01458340
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Proof-of-Concept Study of TD-9855 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Study of TD-9855 in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0085
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2022-03-14 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; ADHD
Keywords: Adult ADHD; Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — ampreloxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TD-9855 Dose 1 (Experimental)
  Interventions: Drug: TD-9855
- Placebo (Experimental)
  Interventions: Drug: Placebo
- TD-9855 Dose 2 (Experimental)
  Interventions: Drug: TD-9855

INTERVENTIONS:
Drug: TD-9855 — Once daily
  Arms: TD-9855 Dose 1
Drug: TD-9855 — Once daily
  Arms: TD-9855 Dose 2
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The safety and efficacy of multiple dosages of TD-9855, administered once daily, will be evaluated in adult males with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following ADHD diagnostic and inclusion criteria:
* Subjects must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for current ADHD subtypes (ADHD combined type, ADHD predominately inattentive type, ADHD predominately hyperactive-impulsive type) as assessed by the clinical interview and confirmed by Adult Attention-Deficit/Hyperactivity Disorder Clinical Diagnostic Scale (ACDS V1.2).
* Subjects must have a total score of 24 or greater on the AISRS at both the Screening and Baseline Visits AND the Baseline Visit AISRS scores must not vary by more than 20% from Screening.
* Subjects are required to have CGI-S score ≥4 (moderate) at both the Screening and Baseline Visits. Subjects should have at least moderate severity for ADHD symptoms.
* For women of childbearing potential, documentation of a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 0. All female subjects of childbearing potential must be using a highly effective method of birth control during the study and for at least 1 month after completion of study drug dosing.
* A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as condom + diaphragm, condom + spermicide, diaphragm + spermicide, or intrauterine device [IUD] with documented failure rate of <1% per year, or oral/injectable/implanted hormonal contraceptives used in combination with a barrier method.
* Women are considered to be not of childbearing potential if they have had a total hysterectomy or bilateral tubal ligation (documentation for either must be provided before enrollment) or are at least 2 years postmenopausal. Female subjects cannot be breast-feeding.

Exclusion Criteria:

Any current psychiatric disorder other than ADHD as defined in DSM-IV-TR as assessed by Mini International Neuropsychiatric Interview (MINI). Subjects with dysthymia that does not require pharmacological treatment will not be excluded.

* MADRS total score >15.
* A diagnosis of ADHD NOS.
* Any diagnosis of lifetime bipolar disorder or psychotic disorder
* A current diagnosis of any severe comorbid Axis II disorder
* Any history of mental retardation, organic mental disorders due to general medical condition or pervasive developmental disorder as defined by DSM-IV-TR.-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 295 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (17):
- United States (17):
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Janus Ctr. for Psychiatric Research, Palm Beach, Florida
  - Carman Research, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Midwest Research Group, Saint Charles, Missouri
  - Ctr. for Psychiatry & Behavioral Med., Las Vegas, Nevada
  - Adult ADHD Program, New York, New York
  - IPS Research, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lincoln Research, Lincoln, Rhode Island
  - CNS Healthcare of Memphis, Memphis, Tennessee
  - FutureSearch Clinical Trials, Austin, Texas
  - Psychiatric & Behavioral Solutions, Salt Lake City, Utah
  - Lifetree Clinical Research, LC, Salt Lake City, Utah
  - Summit Research Network (Seattle), LLC, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Kanodia J, Lo A, Baldwin RM, Graham RA, Bourdet DL. Pharmacokinetics of Ampreloxetine, a Norepinephrine Reuptake Inhibitor, in Healthy Subjects and Adults with Attention-Deficit/Hyperactive Disorder or Fibromyalgia Pain. Clin Pharmacokinet. 2021 Jan;60(1):121-131. doi: 10.1007/s40262-020-00918-7. PMID 32856281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 295 participants with attention-deficit/hyperactivity disorder (ADHD) were enrolled across 19 sites in the United States between December 2011 and September 2013. Participants were randomized in a 1:1:1 ratio, to receive active treatment, consisting of 5 mg or 20 mg of TD-9855 or placebo daily for 6 weeks.
Pre-assignment Details: A total of 295 subjects were randomized into the study and 293 received any amount of study drug.
Groups:
- Placebo: Participants received a matching placebo as oral capsules daily from Day 1 to Day 42.
- TD-9855 5mg: Participants received 5 mg TD-9855 as oral capsules daily from Day 1 to Day 42.
- TD-9855 20 mg: Participants received 10 mg TD-9855 as oral capsules daily from Day 1 to Day 7. Participants' doses were increased to 20 mg from Day 8 to Day 42 based on the safety and tolerability of the 10 mg dose. Participants who in the investigator's opinion were not able to tolerate the 20 mg dose, continued to receive the 10 mg dose from Day 8 to Day 42.
Period: Overall Study
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Started (Intent-to-treat (ITT) population) | 97 | 99 | 99
Received Study Treatment (Safety Analysis Group) | 97 | 98 | 98
Completed | 70 | 78 | 76
Not Completed | 27 | 21 | 23
Not completed — Adverse Event | 5 | 4 | 2
Not completed — Lost to Follow-up | 3 | 3 | 10
Not completed — Miscellaneous | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Protocol Violation | 6 | 6 | 5
Not completed — Withdrawal by Subject | 12 | 6 | 4

BASELINE CHARACTERISTICS:
Population: The ITT population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg | Total
Number analyzed (Participants) | 97 | 99 | 99 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (7.9) | 30.9 (7.4) | 30.5 (7.6) | 30.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 41 | 33 | 104
  Male | 67 | 58 | 66 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 16 | 42
  Not Hispanic or Latino | 84 | 85 | 82 | 251
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 88 | 86 | 84 | 258
  Black or African American | 9 | 9 | 12 | 30
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 1 | 1 | 2
Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score [Mean (Standard Deviation); unit: score on a scale] — A clinician-administered scale that measures all 18 symptoms of adult ADHD using a Likert scale (from 0 [not present] to 3 [severe]). AISRS total score was calculated as sum of all the items on the scale and ranged from 0 to 54.
  score on a scale | 38.4 (7.1) | 39.1 (7.3) | 38.2 (7.1) | 38.6 (7.2)
Barkley Deficits in Executive Functioning Scale - Short Form (BDEFS-SF): Self Report Total Score [Mean (Standard Deviation); unit: score on a scale] — The BDEFS-SF is used to score how frequently the participants experience problems involved in time management; organization and problem solving; self restraint; self motivation; and self-regulation of emotions. The score for each item ranges from 1 (never or rarely) to 4 (very often). The total score on the BDEFS-SF ranges from 20 to 80 with higher scores indicating more frequent problems.
  score on a scale | 52.7 (11.9) | 53.0 (10.5) | 52.3 (10.3) | 52.7 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in AISRS Total Score at Day 42
Description: The AISRS is a modified version of the ADHD Rating Scale that more accurately reflects the impact and severity of ADHD among adults. It is a clinician-administered scale that measures all 18 symptoms of adult ADHD using a Likert scale from 0 (not present) to 3 (severe). The total score ranges from 0 to 54 with a negative change from baseline indicating an improvement in severity/reduction in symptoms.
Time Frame: Baseline and Day 42
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- TD-9855 5mg: Participants received 5 mg TD-9855 as oral capsules once daily from Day 1 to Day 42.
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 97 | 99 | 99
score on a scale | -12.1 (1.21) | -11.7 (1.17) | -12.2 (1.18)
Statistical Analysis 1: Comparison: Placebo vs TD-9855 5mg; Test type: Superiority; p = 0.6026, Mixed Model for Repeated Measures (MMRM) — α=0.05 significance level; One-sided p-values were obtained from the pairwise comparisons between TD-9855 group and placebo group based on the final model; LS Mean Difference = 0.4, 95% CI 1-sided [upper limit 3.2], Standard Error of Mean 1.69
Statistical Analysis 2: Comparison: Placebo vs TD-9855 20 mg; Test type: Superiority; p = 0.4844, MMRM — α=0.05 significance level; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 1-sided [upper limit 2.7], Standard Error of Mean 1.69

2. Secondary Outcome: Change From Baseline in BDEFS-SF: Self Report Total Score at Day 42
Description: The BDEFS-SF: Self-Report is an empirically based tool for evaluating dimensions of adult executive functioning in daily life. The BDEFS-SF is used to score how frequently the participants experience problems involved in time management; organization and problem solving; self restraint; self motivation; and self-regulation of emotions. The score for each item ranges from 1 (never) to 4 (very often). The total score on the BDEFS-SF ranges from 20 to 80 with a negative change from baseline indicating an improvement in functioning.
Time Frame: Baseline and Day 42
Population: The ITT population included all randomized participants. Only participants with data available for analysis and with a with baseline BDEFS-SF Total Score >= 45 are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Participants received matching placebo as oral capsules once per day from Day 1 to Day 42.
- TD-9855 5mg: Participants received 5 mg TD-9855 as oral capsules once per day from Day 1 to Day 42.
- TD-9855 20 mg: Participants received 10 mg TD-9855 as oral capsules once per day from Day 1 to Day 7. Participants' doses were increased to 20 mg from Day 8 to Day 42 based on the safety and tolerability of the 10 mg dose. Participants who in the investigator's opinion were not able to tolerate the 20 mg dose, continued to take the 10 mg from Day 8 to Day 42.
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 75 | 77 | 79
score on a scale | -9.8 (1.56) | -9.7 (1.51) | -11.6 (1.49)
Statistical Analysis 1: Comparison: Placebo vs TD-9855 5mg; Test type: Superiority; p = 0.5269, MMRM — α=0.05 significance level; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.1, 95% CI 1-sided [upper limit 3.7], Standard Error of Mean 2.17
Statistical Analysis 2: Comparison: Placebo vs TD-9855 20 mg; Test type: Superiority; p = 0.2092, MMRM — α=0.05 significance level; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.7, 95% CI 1-sided [upper limit 1.8], Standard Error of Mean 2.16

3. Secondary Outcome: Change From Baseline in AISRS Inattentive Subscale at Day 42
Description: The AISRS is a modified version of the ADHD Rating Scale that more accurately reflects the impact and severity of ADHD among adults. The AISRS inattentive subscale that measures all 9 inattentive symptoms of adult ADHD using a Likert scale from 0 (not present) to 3 (severe). The AISRS inattentive subscale score ranges from 0 to 27 with a negative change from baseline indicating an improvement in severity/reduction in symptoms.
Time Frame: Baseline and Day 42
Population: The ITT population included all randomized participants. Only participants with data available for analysis are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 76 | 82 | 79
score on a scale | -6.2 (6.58) | -6.8 (6.57) | -7.2 (6.72)

4. Secondary Outcome: Change From Baseline in AISRS Hyperactive-impulsive Subscale at Day 42
Description: The AISRS is a modified version of the ADHD Rating Scale that more accurately reflects the impact and severity of ADHD among adults. The AISRS hyperactive-impulsive subscale measures all 9 hyperactive/impulsive symptoms of adult ADHD using a Likert scale from 0 (not present) to 3 (severe). The AISRS hyperactive-impulsive subscale score ranges from 0 to 27 with a negative change from baseline indicating an improvement in severity/reduction in symptoms.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 76 | 82 | 79
score on a scale | -5.2 (5.17) | -5.1 (5.51) | -5.0 (5.11)

5. Secondary Outcome: Percentage of Participants With an AISRS Response at Day 42
Description: The AISRS is a modified version of the ADHD Rating Scale that more accurately reflects the impact and severity of ADHD among adults. The AISRS total scale measures all 18 symptoms of adult ADHD using a Likert scale from 0 (not present) to 3 (severe). The total score ranges from 0 to 54. A responder is defined as a participant with >=30% reduction from baseline in AISRS total score.
Time Frame: Day 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 76 | 82 | 79
percentage of participants | 46.1 | 43.9 | 51.9

6. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score at Day 42
Description: The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participants' illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating 1=normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7,extremely ill. A negative change from baseline indicates a reduction in illness.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 76 | 82 | 79
score on a scale | -1.0 (1.09) | -0.8 (1.13) | -1.0 (1.13)

7. Secondary Outcome: Change From Baseline in Adult ADHD Self-Report Scale (ASRS) Total Score at Day 42
Description: The ASRS is a checklist consisting of the 18 Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV-TR) criteria in which participants rank frequency of each criterion from never (0) to very often (4). The ASRS total score ranges from 0-72 with a negative change from baseline indicating a reduction in frequency of symptoms.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
score on a scale | -12.5 (15.25) | -12.1 (14.49) | -14.0 (13.89)

8. Secondary Outcome: Change From Baseline in ASRS Inattentive Subscale at Day 42
Description: The ASRS inattentive subscale is a checklist consisting of 9 DSM-IV-TR inattentive criteria in which participants rank frequency of each criterion from never (0) to very often (4). The ASRS inattentive subscale score ranges from 0-36 with a negative change from baseline indicating a reduction in frequency of symptoms.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
score on a scale | -6.7 (8.30) | -6.9 (8.26) | -7.7 (7.99)

9. Secondary Outcome: Change From Baseline in ASRS Hyperactive-impulsive Subscale at Day 42
Description: The ASRS hyperactive-impulsive subscale is a checklist consisting of 9 DSM-IV-TR hyperactive/impulsive criteria in which participants rank frequency of each criterion from never (0) to very often (4). The ASRS hyperactive-impulsive subscale score ranges from 0-36 with a negative change from baseline indicating a reduction in frequency of symptoms.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
score on a scale | -5.9 (7.62) | -5.2 (6.94) | -6.3 (6.71)

10. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Day 42
Description: MADRS is a 10-item investigator-rated scale that assesses the range of symptoms that are most frequently observed in patients with major depression. The 10 selected items are rated on a scale of 0 (no depression) to 6 (highest level of depression) with anchors at 2-point intervals. Total scores on the MADRS range from 0 to 60 with a negative change from baseline indicating an improvement in levels of depression.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
score on a scale | -1.3 (3.54) | -0.3 (3.25) | -0.9 (2.86)

11. Secondary Outcome: Percentage of Participants With a Reliable Change on the BDEFS-SF at Day 42
Description: The BDEFS-SF is used to score how frequently the participants experience problems involved in time management; organization and problem solving; self restraint; self motivation; and self-regulation of emotions. The score for each item ranges from 1 (never) to 4 (very often). The total score on the BDEFS-SF ranges from 20 to 80. A reliable change is defined as a decrease in total BDEFS-SF score of 12 or more relative to the baseline value.
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
percentage of participants | 30.4 | 32.6 | 47.6

12. Secondary Outcome: Percentage of Participants With a Reliable Change and Normalized Score on the BDEFS-SF at Day 42
Description: The BDEFS-SF is used to score how frequently the participants experience problems involved in time management; organization and problem solving; self restraint; self motivation; and self-regulation of emotions. The score for each item ranges from 1 (never) to 4 (very often). The total score on the BDEFS-SF ranges from 20 to 80. A reliable change is defined as a decrease in total BDEFS-SF score of 12 or more relative to the baseline value. Normalization is defined as a post-baseline BDEFS-SF total score <45.
Time Frame: Baseline and Day 42
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 62 | 66 | 68
percentage of participants | 29.0 | 28.8 | 38.2

13. Secondary Outcome: Change From Baseline in BDEFS-SF Symptom Count at Day 42
Description: The BDEFS-SF is used to score how frequently the participants experience problems involved in time management; organization and problem solving; self restraint; self motivation; and self-regulation of emotions. A negative change from baseline in symptom count indicates an improvement in functioning. Only symptoms rated as occurring often or very often on the BDEFS-SF are included in the symptom count. Mean change from baseline in symptom count is reported
Time Frame: Baseline and Day 42
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: count of symptoms
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
Number analyzed (Participants) | 79 | 86 | 84
count of symptoms | -3.3 (4.86) | -4.2 (5.72) | -4.5 (5.10)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 56
Description: The Safety Analysis Group included all participants who received study treatment.
Arm/Group | Placebo | TD-9855 5mg | TD-9855 20 mg
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 68/97 | 75/98 | 80/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | TD-9855 5mg (N=98) | TD-9855 20 mg (N=98)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=97) | TD-9855 5mg (N=98) | TD-9855 20 mg (N=98)
Headache (Nervous system disorders) | 17 | 21 | 21
Dizziness (Nervous system disorders) | 9 | 8 | 18
Decreased appetite (Metabolism and nutrition disorders) | 4 | 9 | 13
Fatigue (General disorders) | 6 | 7 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 7 | 10
Insomnia (Psychiatric disorders) | 8 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 2
Middle insomnia (Psychiatric disorders) | 2 | 3 | 6
Nasopharyngitis (Infections and infestations) | 3 | 3 | 5
Nausea (Gastrointestinal disorders) | 2 | 6 | 3
Somnolence (Nervous system disorders) | 6 | 2 | 2
Anxiety (Psychiatric disorders) | 5 | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 1 | 6
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 3 | 4
Tachycardia (Cardiac disorders) | 1 | 2 | 4
Palpitations (Cardiac disorders) | 0 | 2 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 1 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Irritability (General disorders) | 3 | 2 | 2
Feeling jittery (General disorders) | 2 | 1 | 1
Feeling hot (General disorders) | 0 | 3 | 0
Thirst (General disorders) | 1 | 0 | 2
Sluggishness (General disorders) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 4
Blood pressure increased (Investigations) | 1 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood pressure orthostatic increased (Investigations) | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 3 | 3 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 1
Retinal migraine (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 3 | 4
Libido decreased (Psychiatric disorders) | 2 | 2 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 0
Agitation (Nervous system disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Tension (Psychiatric disorders) | 2 | 0 | 0
Anorgasmia (Psychiatric disorders) | 0 | 0 | 1
Apathy (Psychiatric disorders) | 0 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Derealisation (Psychiatric disorders) | 0 | 1 | 0
Elevated mood (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Terminal insomnia (Psychiatric disorders) | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 1 | 0
Liposuction (Surgical and medical procedures) | 0 | 0 | 1
Mammoplasty (Surgical and medical procedures) | 0 | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 4 | 0
Flushing (Vascular disorders) | 0 | 0 | 2
Hot flush (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No